CLINICAL TRIAL: NCT01483963
Title: A Phase 2a, Open-label, Dose-ranging Study of the Safety and Effectiveness of AA4500 for the Treatment of Adhesive Capsulitis of the Shoulder
Brief Title: AA4500 for the Treatment of Adhesive Capsulitis of the Shoulder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUX-CC-870
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Adhesive Capsulitis; Frozen Shoulder
MeSH Terms: conditions — Bursitis | interventions — Microbial Collagenase; xiapex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- AA4500 0.29 mg/1 mL (Experimental): Up to three injections
  Interventions: Biological: AA4500 0.29 mg/1 mL; Other: Shoulder exercises
- AA4500 0.58 mg/2 mL (Experimental): Up to three injections
  Interventions: Biological: AA4500 0.58 mg/2 mL; Other: Shoulder exercises
- AA4500 0.58 mg/1 mL (Experimental): Up to three injections
  Interventions: Biological: AA4500 0.58 mg/1 mL; Other: Shoulder exercises
- AA4500 0.58 mg/0.5 mL (Experimental): Up to three injections
  Interventions: Biological: AA4500 0.58 mg/0.5 mL; Other: Shoulder exercises
- Shoulder exercises (Other): Home shoulder exercises for 64 days
  Interventions: Other: Shoulder exercises

INTERVENTIONS:
Biological: AA4500 0.29 mg/1 mL — treatment of adhesive capsulitis
  Other Names: collagenase clostridium histolyticum; XIAFLEX; XIAPEX
  Arms: AA4500 0.29 mg/1 mL
Biological: AA4500 0.58 mg/2 mL — treatment of adhesive capsulitis
  Other Names: collagenase clostridium histolyticum; XIAFLEX; XIAPEX
  Arms: AA4500 0.58 mg/2 mL
Biological: AA4500 0.58 mg/1 mL — treatment of adhesive capsulitis
  Other Names: collagenase clostridium histolyticum; XIAFLEX; XIAPEX
  Arms: AA4500 0.58 mg/1 mL
Biological: AA4500 0.58 mg/0.5 mL — treatment of adhesive capsulitis
  Other Names: collagenase clostridium histolyticum; XIAFLEX; XIAPEX
  Arms: AA4500 0.58 mg/0.5 mL
Other: Shoulder exercises — Home shoulder exercises, minimum of 3 times per day

SUMMARY:
The objectives of this study are to assess the safety, effectiveness, and immunogenicity of AA4500 in the treatment of adhesive capsulitis.

DETAILED DESCRIPTION:
This study is a Phase 2a, open-label, dose-ranging study of the safety and effectiveness of AA4500 for the treatment of adhesive capsulitis of the shoulder. To be eligible for treatment, a subject must have unilateral idiopathic adhesive capsulitis of the shoulder with restricted range of motion in the affected shoulder for at least 3 months but not more than 12 months. Subjects will be screened for study eligibility within 30 days before injection of study drug.

Approximately 50 adult women and men are to be enrolled in this study. Following screening and determination of study eligibility, Assignment to Cohorts 1-4 is sequential. Subjects assigned to Cohorts 1 through 4 may receive up to 3 injections of AA4500 according to cohort assignment. Each injection will be separated by a minimum of 21 days. Subjects assigned to Cohort 5 will receive home shoulder exercises only, while subjects assigned to Cohorts 1-4 will receive AA4500 and home shoulder exercises. Subjects in Cohort 5 will be offered physical therapy sessions for a period of 2 months following completion of the study.

Dosing will range from 0.29 mg to 0.58 mg with varying volumes.

ELIGIBILITY:
Inclusion Criteria:

1. Be a male or female and be greater than or equal to 18 years of age
2. If a female of childbearing potential, have a negative urine pregnancy test and be using an effective contraception method (ie, abstinence, intrauterine device (IUD), hormonal (estrogen/progestin) contraceptives, or barrier control) for at least one menstrual cycle prior to study enrollment and for one menstrual cycle following end of study, or be surgically sterile
3. Have unilateral idiopathic adhesive capsulitis of one shoulder for at least 3 months but not more than 12 months before the screening visit and be in Stage 2 (frozen or adhesive stage), as determined by the investigator
4. Have normal range of motion in the contralateral shoulder, as determined by the investigator
5. Have restricted active range of motion (AROM) in the affected shoulder defined as: a deficit of at least 60 degrees in total AROM in the affected shoulder as compared with the total AROM in the contralateral shoulder and a deficit of at least 30 degrees in AROM in at least one of the following planes as compared with the contralateral shoulder:

   * Forward flexion
   * Abduction
   * External rotation with the elbow up to 90 degrees abduction
   * Internal rotation with the elbow up to 90 degrees abduction
6. Voluntarily sign and date an informed consent agreement approved by the Institutional Review Board/Independent Ethics Committee (IRB/IEC). The subject must also sign an authorization form to allow disclosure of his protected health information (PHI). The PHI authorization form and informed consent form may be an integrated form or may be separate forms depending on the institution.
7. Be able to complete and understand the various rating instruments in English.

Exclusion Criteria:

1. Is a pregnant or lactating female or female intending to become pregnant during the study
2. Is a male who intends to father a child during the study
3. Has received treatment for adhesive capsulitis or is planning to receive treatment for adhesive capsulitis at any time during the study including but not limited to:

   * physical therapy or acupuncture within 2 weeks before the first injection of AA4500
   * intra-articular or intrabursal injection(s) of lidocaine; suprascapular nerve blocks; corticosteroids; electroanalgesic and/or thermoanalgesic modalities within 1 month before the screening visit
   * intra-articular or intrabursal injection(s) of sodium hyaluronate within 3 months before the screening visit
   * glenohumeral distension arthrography and/or surgical intervention (including shoulder manipulation under anesthesia) at any time
4. Has any of the following conditions, as determined by the investigator:

   * Adhesive capsulitis as a result of traumatic injury
   * Pain in the affected shoulder at rest that is greater than or equal to 4 on the 11-point pain scale
   * Active subacromial impingement in the affected shoulder
   * Calcified tendonitis in the affected shoulder
   * Glenohumeral joint arthritis in the affected shoulder
   * Arthrosis of the affected shoulder
   * Chondrolysis of the affected shoulder
   * Subscapularis tendon rupture of the affected shoulder
   * Other rotator cuff injuries of the affected shoulder
   * Uncontrolled hypertension
   * Uncontrolled diabetes
   * Uncontrolled thyroid disease
   * History of thrombosis or post-thrombosis syndrome
   * Physical impairment that would preclude performing the protocol defined exercises
   * Active infection in area to be treated
   * Clinically significant neurological disease
   * Coagulation disorder, using anticoagulant (except for less than or equal to 150 mg aspirin) within 7 days prior to each injection day
   * Known active hepatitis B or C (history of hepatitis A permitted)
   * Other significant medical condition (eg, morbid obesity, cervical disc disease), which in the investigator's opinion would make the subject unsuitable for enrollment in the study
5. Is unwilling or unable to cooperate with the requirements of the study including completion of all scheduled study visits.
6. Has received oral or intravenous steroids for any reason within 3 weeks before the screening visit
7. Has received an investigational drug or treatment within 30 days before the first dose of study drug.
8. Has a known systemic allergy to collagenase or any other excipient of AA4500 or any other procedural medication.
9. Has, at any time, received collagenase for the treatment of adhesive capsulitis.
10. Is unable to undergo an x-ray or MRI (contraindication) evaluation of the affected shoulder.
11. Is planning to be treated with commercial Xiaflex at any time during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil H Shusterman, MD FACP, Study Director — Endo Pharmaceuticals
Locations (15):
- United States (15):
  - Alabama Orthopaedic Center - Research, Birmingham, Alabama
  - HOPE Research Institute, Phoenix, Arizona
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - OrthoArkansas, Little Rock, Arkansas
  - CORE Orthopaedic Medical Center, Encinitas, California
  - Triwest Research Associates, La Mesa, California
  - Advent Clinical Research, Pinellas Park, Florida
  - Rockford Orthopedic Associates, Rockford, Illinois
  - The Indiana Hand to Shoulder Center, Indianapolis, Indiana
  - Stony Brook University Medical Center, Stony Brook, New York
  - David R. Mandel, MD, Inc., Cleveland, Ohio
  - Health Research Institute, Oklahoma City, Oklahoma
  - Blair Orthopedic Associates, Inc., Altoona, Pennsylvania
  - Alpha Clinical Research, LLC, Clarksville, Tennessee
  - Basin Orthopedic Surgical Specialists, Odessa, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- AA4500 0.29 mg/1 mL: Up to 3 injections of collagenase clostridium histolyticum (AA4500) 0.29 mg/1 mL
  Shoulder exercises: Home shoulder exercises, minimum of 3 times per day
- AA4500 0.58 mg/2 mL: Up to 3 injections of AA4500 0.58 mg/2 mL
  Shoulder exercises: Home shoulder exercises, minimum of 3 times per day
- AA4500 0.58 mg/1 mL: Up to 3 injections of AA4500 0.58 mg/1 mL
  Shoulder exercises: Home shoulder exercises, minimum of 3 times per day
- AA4500 0.58 mg/0.5 mL: Up to 3 injections of AA4500 0.58 mg/0.5 mL
  Shoulder exercises: Home shoulder exercises, minimum of 3 times per day
- Shoulder Exercises Only: Home shoulder exercises for 64 days
  Shoulder exercises: Home shoulder exercises, minimum of 3 times per day
Period: Overall Study
Arm/Group | AA4500 0.29 mg/1 mL | AA4500 0.58 mg/2 mL | AA4500 0.58 mg/1 mL | AA4500 0.58 mg/0.5 mL | Shoulder Exercises Only
Started | 10 | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AA4500 0.29 mg/1 mL: Up to 3 injections of AA4500 0.29 mg/1 mL
  Shoulder exercises: Home shoulder exercises, minimum of 3 times per day
- Total: Total of all reporting groups
Arm/Group | AA4500 0.29 mg/1 mL | AA4500 0.58 mg/2 mL | AA4500 0.58 mg/1 mL | AA4500 0.58 mg/0.5 mL | Shoulder Exercises Only | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (4.93) | 54.1 (8.81) | 58.4 (8.97) | 53.2 (5.71) | 55.1 (7.02) | 54.0 (7.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 9 | 8 | 7 | 40
  Male | 2 | 2 | 1 | 2 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 8 | 10 | 10 | 10 | 10 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 9 | 10 | 9 | 10 | 10 | 48
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 10 | 10 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 92 in Active Forward Flexion
Description: Active range of motion (AROM) measurement using a goniometer to assess forward flexion in the affected shoulder
Time Frame: Baseline, Day 92
Population: All participants who have a baseline AROM measurement of the affected shoulder and at least 1 measurement of AROM of the affected shoulder following the first administration of study drug (AA4500 groups) or post baseline (shoulder exercises only group)
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | AA4500 0.29 mg/1 mL | AA4500 0.58 mg/2 mL | AA4500 0.58 mg/1 mL | AA4500 0.58 mg/0.5 mL | Shoulder Exercises Only
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
degrees | 22.9 (13.83) | 37.5 (22.89) | 42.9 (30.64) | 23.8 (41.97) | 12.0 (12.68)

2. Secondary Outcome: Change From Baseline to Day 92 in Passive Forward Flexion
Description: Passive range of motion (PROM) measurement using a goniometer to assess forward flexion in the affected shoulder
Time Frame: Baseline, Day 92
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | AA4500 0.29 mg/1 mL | AA4500 0.58 mg/2 mL | AA4500 0.58 mg/1 mL | AA4500 0.58 mg/0.5 mL | Shoulder Exercises Only
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
degrees | 21.8 (11.92) | 39.1 (22.13) | 46.2 (20.35) | 10.5 (23.96) | 12.0 (14.13)

3. Secondary Outcome: Change From Baseline to Day 92 in Active Abduction
Description: AROM measurement using a goniometer to assess abduction in the affected shoulder
Time Frame: Baseline, Day 92
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | AA4500 0.29 mg/1 mL | AA4500 0.58 mg/2 mL | AA4500 0.58 mg/1 mL | AA4500 0.58 mg/0.5 mL | Shoulder Exercises Only
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
degrees | 28.4 (15.81) | 36.0 (32.94) | 53.7 (27.59) | 35.8 (41.02) | 16.7 (8.06)

4. Secondary Outcome: Change From Baseline to Day 92 in Passive Abduction
Description: PROM measurement using a goniometer to assess abduction in the affected shoulder
Time Frame: Baseline, Day 92
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | AA4500 0.29 mg/1 mL | AA4500 0.58 mg/2 mL | AA4500 0.58 mg/1 mL | AA4500 0.58 mg/0.5 mL | Shoulder Exercises Only
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
degrees | 28.6 (15.69) | 44.8 (34.69) | 56.1 (30.05) | 18.0 (40.87) | 24.3 (29.69)

5. Secondary Outcome: Change From Baseline to Day 92 in Active External Rotation
Description: AROM measurement using a goniometer to assess external rotation in the affected shoulder
Time Frame: Baseline, Day 92
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | AA4500 0.29 mg/1 mL | AA4500 0.58 mg/2 mL | AA4500 0.58 mg/1 mL | AA4500 0.58 mg/0.5 mL | Shoulder Exercises Only
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
degrees | 24.8 (13.39) | 19.7 (27.49) | 16.6 (16.79) | 7.4 (29.15) | 6.0 (27.87)

6. Secondary Outcome: Change From Baseline to Day 92 in Passive External Rotation
Description: PROM measurement using a goniometer to assess external rotation in the affected shoulder
Time Frame: Baseline, Day 92
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | AA4500 0.29 mg/1 mL | AA4500 0.58 mg/2 mL | AA4500 0.58 mg/1 mL | AA4500 0.58 mg/0.5 mL | Shoulder Exercises Only
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
degrees | 20.0 (9.64) | 19.3 (24.57) | 40.9 (33.71) | 9.1 (29.32) | 10.7 (20.27)

7. Secondary Outcome: Change From Baseline to Day 92 in Active Internal Rotation
Description: AROM measurement using a goniometer to assess internal rotation with the elbow up to 90° abduction in the affected shoulder
Time Frame: Baseline, Day 92
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | AA4500 0.29 mg/1 mL | AA4500 0.58 mg/2 mL | AA4500 0.58 mg/1 mL | AA4500 0.58 mg/0.5 mL | Shoulder Exercises Only
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
degrees | 8.1 (14.12) | 13.0 (20.85) | 9.5 (26.87) | 17.4 (24.43) | 1.2 (20.92)

8. Secondary Outcome: Change From Baseline to Day 92 in Passive Internal Rotation
Description: PROM measurement using a goniometer to assess internal rotation with the elbow up to 90° abduction in the affected shoulder
Time Frame: Baseline, Day 92
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | AA4500 0.29 mg/1 mL | AA4500 0.58 mg/2 mL | AA4500 0.58 mg/1 mL | AA4500 0.58 mg/0.5 mL | Shoulder Exercises Only
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
degrees | 8.4 (16.87) | 19.8 (21.70) | 13.1 (23.38) | 23.6 (18.77) | 2.9 (17.55)

9. Secondary Outcome: Change From Baseline to Day 92 in American Shoulder and Elbow Surgeons (ASES) Composite Score
Description: Composite score ranging from 0-100, with 0 being worst pain and function loss, derived from the sum of the scores from pain subscale (11-point NRS where 0=no pain at all and 10=pain) and function subscale (activity questionnaire where 0=unable to do to, 1=very difficult to do, 2=somewhat difficult, and 3=not difficult); adapted from ASES Standardized Shoulder Assessment Form, Patient Self-Evaluation
Time Frame: Baseline, Day 92
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 0.29 mg/1 mL | AA4500 0.58 mg/2 mL | AA4500 0.58 mg/1 mL | AA4500 0.58 mg/0.5 mL | Shoulder Exercises Only
Number analyzed (Participants) | 10 | 9 | 9 | 10 | 10
units on a scale | 26.9 (13.17) | 41.6 (18.99) | 35.9 (24.33) | 19.3 (24.29) | 9.9 (15.84)

10. Secondary Outcome: Change From Baseline to Day 92 in ASES Pain Subscale
Description: Pain subscale score ranging from 0-50, with 0 being greatest pain, derived from participant assessment of pain in response to "How bad is the pain in your affected shoulder today?" on an 11-point numerical rating scale (NRS) where 0=no pain at all and 10=pain as bad as it can be and calculated as (10 - NRS score) x 5); adapted from ASES Standardized Shoulder Assessment Form, Patient Self-Evaluation
Time Frame: Baseline, Day 92
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 0.29 mg/1 mL | AA4500 0.58 mg/2 mL | AA4500 0.58 mg/1 mL | AA4500 0.58 mg/0.5 mL | Shoulder Exercises Only
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
units on a scale | 10.0 (11.06) | 15.5 (13.22) | 15.5 (14.99) | 8.0 (12.52) | 1.5 (11.32)

11. Secondary Outcome: Change From Baseline to Day 92 in ASES Function Subscale
Description: Function subscale score ranging from 0-50, with 0 being most dysfunctional, derived from participant assessment of ability to do 10 activities with affected shoulder/arm where 0=unable to do to, 1=very difficult to do, 2=somewhat difficult, and 3=not difficult, and calculated as (cumulative total score for the 10 activity items) × (5/3); adapted from ASES Standardized Shoulder Assessment Form, Patient Self-Evaluation
Time Frame: Baseline, Day 92
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 0.29 mg/1 mL | AA4500 0.58 mg/2 mL | AA4500 0.58 mg/1 mL | AA4500 0.58 mg/0.5 mL | Shoulder Exercises Only
Number analyzed (Participants) | 10 | 10 | 9 | 9 | 10
units on a scale | 17.4 (8.72) | 26.0 (10.98) | 19.2 (12.36) | 11.3 (13.53) | 8.4 (5.85)

12. Secondary Outcome: Subject Satisfaction With Treatment at Day 92
Description: Participant assessment of satisfaction with treatment rated as very satisfied, quite satisfied, neither satisfied nor dissatisfied, quite dissatisfied, or very dissatisfied.
Time Frame: Day 92
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AA4500 0.29 mg/1 mL | AA4500 0.58 mg/2 mL | AA4500 0.58 mg/1 mL | AA4500 0.58 mg/0.5 mL | Shoulder Exercises Only
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  Very satisfied | 4 | 6 | 8 | 3 | 5
  Quite satisfied | 4 | 2 | 1 | 3 | 2
  Neither satisfied nor dissatisfied | 2 | 1 | 0 | 3 | 3
  Quite dissatisfies | 0 | 1 | 1 | 1 | 0
  Very dissatisfied | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Investigator Assessment of Improvement With Treatment at Day 92
Description: Investigator assessment of degree of improvement in severity of the participant's treated shoulder compared with screening rated as very much improved, much improved, minimally improved, no change, minimally worse, much worse, or very much worse.
Time Frame: Day 92
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AA4500 0.29 mg/1 mL | AA4500 0.58 mg/2 mL | AA4500 0.58 mg/1 mL | AA4500 0.58 mg/0.5 mL | Shoulder Exercises Only
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  Very much improved | 1 | 5 | 7 | 3 | 2
  Much improved | 3 | 2 | 2 | 1 | 2
  Minimally improved | 5 | 2 | 1 | 5 | 3
  No change | 1 | 0 | 0 | 1 | 2
  Minimally worse | 0 | 1 | 0 | 0 | 1
  Much worse | 0 | 0 | 0 | 0 | 0
  Very much worse | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 129 days (up to 30 day screening period and 92±7 day study period)
Arm/Group | AA4500 0.29 mg/1 mL | AA4500 0.58 mg/2 mL | AA4500 0.58 mg/1 mL | AA4500 0.58 mg/0.5 mL | Shoulder Exercises Only
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/10 | 9/10 | 10/10 | 10/10 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 0.29 mg/1 mL (N=10) | AA4500 0.58 mg/2 mL (N=10) | AA4500 0.58 mg/1 mL (N=10) | AA4500 0.58 mg/0.5 mL (N=10) | Shoulder Exercises Only (N=10)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 1 (2) | 1 (3) | 0 (0) | 0 (0)
Injection site coldness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 4 (7) | 4 (7) | 3 (4) | 6 (8) | 0 (0)
Injection site haemorrhage (General disorders) | 1 (1) | 2 (4) | 3 (4) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 6 (11) | 6 (13) | 6 (14) | 4 (6) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 2 (2) | 3 (3) | 2 (3) | 5 (6) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accident at work (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 4 (7) | 2 (2) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Hypokinesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes